CLINICAL TRIAL: NCT03454789
Title: Comparison of the Onset Times and Durations of Actions of Different Local Anesthetic Mixture Solutions Used for Ultrasound-guided Axillary-supraclavicular Brachial Plexus Blocks for Upper Limb Trauma Surgery
Brief Title: Comparison of the Onset Times and Durations of Actions of Different Local Anesthetic Mixture Solutions [CODLAM]
Acronym: CODLAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Collaborators: Medical University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 6940
Record Dates: First submitted 2018-02-16; First posted 2018-03-06 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Injury Arm
Keywords: brachial plexus block; local anesthetic mixture solution; axillary-supraclavicular approach; outcome quality; lidocaine, bupivacaine; onset time; duration action local anesthetic; postoperative analgesia
MeSH Terms: conditions — Arm Injuries | interventions — Brachial Plexus Block

STUDY DESIGN:
Intervention Model Description: LB= 15 ml lidocaine 1% + 15 ml bupivacaine 0.5%; BS= 20 ml bupivacaine 0.5% + 10 ml normal saline; LS=20 ml lidocaine 1% + 10 ml normal saline; and BL=20 ml bupivacaine 0.5% + 10 ml lidocaine 1%.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, the operating team, nurses, and observers involved in the quality assessment of blocks and the follow-up data collection were unaware of group allocation. The research coordinator after the BPB was not present in the operating theatre at the time of tourniquet inflation and the beginning of the surgery. The intra- and postoperative parameters, drug consumptions and VNR values were collected and matched retrospectively, the list of cases was provided in the form of a spreadsheet program by an observer-blinded assistant and was statistically evaluated by an independent analyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LB Group (Active Comparator): Ultrasound-guided brachial plexus block for LB Group (15 ml lidocaine 1% + 15 ml bupivacaine 0.5%)
  Interventions: Drug: brachial plexus block for LB Group
- BS Group (Active Comparator): Ultrasound-guided brachial plexus block for BS Group (20 ml bupivacaine 0.5% + 10 ml normal saline)
  Interventions: Drug: brachial plexus block for BS Group
- LS Group (Active Comparator): Ultrasound-guided brachial plexus block for LS Group (20 ml lidocaine 1% + 10 ml normal saline)
  Interventions: Drug: brachial plexus block for LS Group
- BL Group (Active Comparator): and Ultrasound-guided brachial plexus block for BL Group (20 ml bupivacaine 0.5% + 10 ml lidocaine 1%)
  Interventions: Drug: brachial plexus block for BL Group

INTERVENTIONS:
Drug: brachial plexus block for LB Group — Standardized UG AX-SC approach to the BP was performed under sterile conditions by the same anesthesiologist. SC block was performed with the traditional in-plane, single injection cluster approach, then AX approach was performed in the supine position, with a standardized dose of 0.4 ml/kg BW
  Other Names: Lidocain-Egis 1% Bucain Actavis 5 mg/ml,1:1
  Arms: LB Group
Drug: brachial plexus block for BS Group — Standardized UG AX-SC approach to the BP was performed under sterile conditions by the same anesthesiologist. SC block was performed with the traditional in-plane, single injection cluster approach, then AX approach was performed in the supine position, with a standardized dose of 0.4 ml/kg BW
  Other Names: Bucain Actavis 5 mg /ml
  Arms: BS Group
Drug: brachial plexus block for LS Group — Standardized UG AX-SC approach to the BP was performed under sterile conditions by the same anesthesiologist. SC block was performed with the traditional in-plane, single injection cluster approach, then AX approach was performed in the supine position, with a standardized dose of 0.4 ml/kg BW
  Other Names: Lidocain Egis 1%
  Arms: LS Group
Drug: brachial plexus block for BL Group — Standardized UG AX-SC approach to the BP was performed under sterile conditions by the same anesthesiologist. SC block was performed with the traditional in-plane, single injection cluster approach, then AX approach was performed in the supine position, with a standardized dose of 0.4 ml/kg BW
  Other Names: Bucain Actavis 5 mg/ml, Lidocain-Egis 1% 2:1
  Arms: BL Group

SUMMARY:
Objective To investigate the onset times and duration of local anesthetic mixture solutions used for axillary-supraclavicular brachial plexus blocks and to compare the quality of anesthesia in patients with trauma of the upper limb.

Design Randomized-prospective, observational study. Setting Perioperative, Trauma Clinic, University of Pecs, Hungary. Participants 85 consecutive, unpremedicated ASA physical status I-III patients, between the ages of 19 and 83, scheduled for trauma surgery of the hand and forearm.

Interventions Patients assigned to four groups for standardized ultrasound guided axillary-supraclavicular block with lidocaine 1% and bupivacaine 0,5% 1:1 mixture (Group LB, n = 17) or bupivacaine 0.33% (Group BS, n = 14) or lidocaine 0,66% (Group LS, n = 14) or bupivacaine 0.5% and lidocaine 1% 2:1 mixture (Group BL, n = 40). Total target volume of 0.4 ml/kg was administered to both groups.

Measurements Data were collected on patient demographics, the onset times and the duration of actions of local anesthetic mixtures were measured, the tourniquet discomfort, vital parameters, pre and postoperative verbal numeric rating scale of pain intensity, anxiolytic/analgesic consumption and the complications were recorded. The quality of anesthesia was assessed by a sensory-motor-coping-pain scale (0-16).

DETAILED DESCRIPTION:
Total of 93 American Society of Anesthesiologist (ASA) I-III consecutive adult patients aged between 19 and 83 years old scheduled for elective or emergency trauma surgery of hand and forearm under ultrasound-guided brachial plexus block (UG BPB) between 17.01. and 15.08. in 2017 were assigned to this randomized-prospective observational study after approval by the University Research Ethics Board. Patients were excluded if continuous peripheral nerve catheter technique or bilateral block was planned, or the patient refused to participate. Exclusion criteria included psycho-mental conditions interfering with consent or assessment; pre-existing chronic pain condition or daily analgesic or sedative consumption; sedative or analgesic premedication; pre-existing neurological disorders aﬀecting the brachial plexus (BP); obstructive sleep apnea; contraindications to BPB including local skin infections or allergy to local anesthetic (LA) agents. After exclusion, eligible patients for the study were randomized to four LA mixture solution groups and analyzed and presented in a Consolidated Standards of Reporting Trials flow diagram. Standardized UG axillary-supraclavicular (AX-SC) approach to the BP was performed under sterile conditions by the same anesthesiologist. The standardized dose was 0.4 ml/kg, the targeted maximized single shot volume was 30 ml. After administration of LA, standard anesthesia monitoring was started in the operating room. Data were collected as baseline (T0); intraoperative mean values (Top); postoperative values straight after surgery (Tpop); 6 and 24 after surgery (T6; T24) including measurement of heart rate (HR), non-invasive arterial blood pressure (NIBP), and verbal numeric rate (VNR, 11 point scale) of pain intensity. The extent of sensory and motor blockade was assessed meticulously in the corresponding region after the total dose of LA was injected until the blockade was defined as completed. Sensory block was tested by pinching and touching the skin of the arm and hand at the areas innervated by the four nerves. A von Frey filament with a standard target force of 10 gr (Touch Test ® Sensory Evaluator, Red 5,07; USA) was used for the assessment of the loss of protective sensation. The outcome quality and success rate of BPB was assessed by a composite tool designed for evaluating the loss of sensory (S, 0-4: failed to excellent), motor function (M, 0-4: failed to excellent), the coping of the patient (C, 0-4: failed to excellent) and the postoperative pain at the end of surgery and 24 h after (P, 0-4: pain before the end of surgery to long-lasting - 24 h - analgesia). The overall quality of PNB was evaluated by independent examiners, based on the aggregate 0-16 point scale. Under 7 Point the block was defined as failed, 8-11 = Tolerable; 12-13 = Good; 14-16 = Excellent. The duration of anesthesia was defined as the time between the end of the LA injection for BPB and the return of the sensory function reported by the patient or the necessity for first analgesic medication.

The study was conducted comparing the onset times and the duration of sensory effects of the same volumes of lidocaine-bupivacaine 1:1 mixture (LB), bupivacaine in normal saline (BS), lidocaine in normal saline (LS), and bupivacaine-lidocaine 2:1 mixture (BL) for BPB. Midazolam and fentanyl consumption were analyzed in the four groups, the outcome quality of blocks, vital parameters, visual numeric rate (VNR) of pain intensity values and non-steroid analgesic consumptions were compared between the four groups.

The IBM SPSS Statistics (Windows, version 24, 2016) was used in our analyses. Paired samples t-test, Kruskal-Wallis test combined with the Mann-Whitney U test for post hoc testing were used in analyzing the ordinal data. The Chi-square test was used for comparison of the categorical variables between the groups. ANOVA combined with Bonferroni post hoc test was used in analyzing the variance of linear data between groups. P<0.05 was considered significant.

Priori power calculation was performed by GPower 3.1.9.2 version: effect size f=0.4, alfa err=0.05; power=0.85; number of groups=4; total sample size=84.

ELIGIBILITY:
Inclusion Criteria:

* elective or emergency trauma surgery of hand or forearm
* consented to ultrasound-guided BPB

Exclusion Criteria:

* continuous peripheral nerve catheter technique or bilateral block was planned
* the patient refused to participate
* psycho-mental conditions interfering with consent or assessment
* pre-existing chronic pain condition or daily analgesic or sedative consumption
* sedative or analgesic premedication
* pre-existing neurological disorders aﬀecting the brachial plexus
* obstructive sleep apnea
* contraindications to PNB including local skin infections or allergy to LA agents.

Ages: 19 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
onset time | 0-30 minutes
  Complete sensory block was defined by loss of sensation of filament prick and touch on all four nerve distribution. Complete motor block was defined by the loss of thumb abduction, thumb adduction, thumb opposition, and flexion at elbow.

SECONDARY OUTCOMES:
duration of action | 1-22 hours
  The duration of anesthesia was defined as the time between the end of the LA injection for BPB and the return of the sensory function reported by the patient or the necessity for first analgesic medication.
The outcome quality of BPB. | 24-48 hours
  The outcome quality was assessed by a composite tool designed for evaluating the loss of sensory (S, 0-4: failed to excellent), motor function (M, 0-4: failed to excellent), the coping of the patient (C , 0-4: failed to excellent) and the postoperative pain at the end of surgery and 24 h after (P, 0-4: pain before the end of surgery to long-lasting - 24 h - analgesia).
Success rate of BPB. | 3-14 days
  The rate of Excellent, Good, Tolerable and Failed in the four groups. The overall quality of PNB was evaluated by independent examiners, based on the aggregate 0-16 point scale. Under 7 Point the block was defined as failed, 8-11 = Tolerable; 12-13 = Good; 14-16 = Excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Lajos Bogar, Prof, Study Director — Department of Anesth.and Int Care,University of Pecs, Medical School

IPD SHARING:
Plan to Share IPD: Undecided